CLINICAL TRIAL: NCT06451380
Title: Patient-controlled Sedation With Propofol Versus Anesthesiologist-administered Sedation for Orthopedic Surgery Under Regional Anesthesia : a Prospective Randomized Trial
Brief Title: Patient-controlled Sedation With Propofol Versus Anesthesiologist-administered Sedation for Orthopedic Surgery
Acronym: PACOSA
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: GCS Ramsay Santé pour l'Enseignement et la Recherche (Other)
Collaborators: Euraxi Pharma (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2024-A00628-39
Record Dates: First submitted 2024-06-04; First posted 2024-06-11 (Actual); Last update posted 2025-11-24 (Actual); Status verified 2025-11

CONDITIONS: Orthopedic Disorder
MeSH Terms: conditions — Musculoskeletal Diseases

STUDY DESIGN:
Intervention Model Description: This is an interventional, prospective, randomized, open-label, controlled, single-center study.
Masking Description: This is a randomized, open-label study.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Patient-controlled propofol sedation (Experimental): Patients in the experimental arm will receive self-controlled sedation using a programmable infusion device, which will deliver boluses of propofol at the patient's request.
  The initial dose of propofol, the bolus dose and the refractory period will be determined according to a standardized protocol used in current practice.
  Patients will be trained in the use of the device prior to the procedure. An anesthetist will be present to monitor the patient and intervene in the event of complications.
  Interventions: Procedure: orthopaedic surgery; Drug: propofol anesthesia
- Anesthesiologist-controlled propofol sedation (Active Comparator): Patients in the control arm will receive sedation administered and monitored by an anesthetist, who will adjust the dose of propofol according to the patient's needs.
  A standardized protocol for propofol administration and dose adjustment criteria will be followed until a mild sedation score is achieved.
  The anesthetist will continuously monitor the patient and adjust the sedation accordingly.
  Interventions: Procedure: orthopaedic surgery; Drug: propofol anesthesia

INTERVENTIONS:
Procedure: orthopaedic surgery — orthopaedic surgery of the upper limb under anaesthesia
Drug: propofol anesthesia — The initial dose of propofol and the refractory period will be determined according to a standardized protocol used in current practice.

SUMMARY:
The purpose of this study is to compare patient satisfaction with patient-controlled sedation with propofol and anesthesiologist-controlled sedation during orthopedic procedures of the upper limb under locoregional anesthesia.

DETAILED DESCRIPTION:
This is an interventional, prospective, randomized, open-label, controlled, single-center study designed to evaluate the less commonly used patient-controlled sedation, comparing it with sedation administered by the anesthesiologist in a population of patients indicated for orthopedic upper limb surgery requiring additional sedation.

Once informed consent has been signed, patients will be randomized into one of two study arms in a 1:1 ratio, stratified by age:

* Experimental arm (1) : patient-controlled propofol sedation ;
* Control arm (2) : anesthesiologist-controlled propofol sedation.

Patient participation in the study lasts from 1 to 7 days maximum (from preoperative inclusion to hospital discharge).

ELIGIBILITY:
Inclusion Criteria:

* Patients aged 18 and over;
* Patients indicated for orthopedic surgery of the upper limb under anaesthesia requiring additional sedation;
* Ability to use the patient-controlled sedation device;
* Body Mass Index less than 40 kg/m²;
* American Society of Anesthesiologists Class I to III;
* Patient agreeing to study assessments and follow-up visits
* Patient having been informed and agreeing to participate in the study by signing an informed consent form.

Exclusion Criteria:

* Contraindications to locoregional anesthesia (allergy, local infection, coagulation disorders);
* Surgery of the upper limb not compatible with locoregional anesthesia (arthroplasty);
* Patient unable to understand study information for linguistic, psychological or cognitive reasons linguistic, psychological or cognitive reasons ;
* Patient pregnant or likely to be pregnant, of childbearing age, without effective contraception or breastfeeding ;
* Patient participating in another clinical trial, or in a period of exclusion from another clinical trial;
* Patient under legal protection, or deprived of liberty by judicial or administrative decision administrative ;
* Patient not covered by a social security scheme.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 70 (Actual)
Dates: Start 2024-10-02 (Actual); Primary Completion 2025-01-09 (Actual); Study Completion 2025-01-09 (Actual)

PRIMARY OUTCOMES:
patient satisfaction | up to 7 days
  Comparison between the 2 groups of patient satisfaction assessed by the total score of the Evaluation of the Experience of Locoregional Anesthesia at the end of the procedure, once the patients had left the recovery room.

CONTACTS AND LOCATIONS:
Locations (1):
- Clinique Jouvenet, Paris, France